CLINICAL TRIAL: NCT05602688
Title: Study to Investigate Melissa Officinalis L. Supplementation for Emotional Health and Sleep Disturbance: A Perspective, Randomized, Double-blinded, Placebo-controlled, Parallel-group Clinical Trial
Brief Title: Melissa Officinalis L. Supplementation for Emotional Health and Sleep Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayub Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RC-2022/EA-01/194
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Depression; Anxiety; Stress; Insomnia
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Experimental): This arm will receive oral 200 mg Lemon Balm supplement tablet two times a day for three-weeks.
  Interventions: Dietary Supplement: Lemon Balm Supplement
- Control group (Active Comparator): This arm will receive an oral matched placebo tablet two times a day for three-weeks.
  Interventions: Dietary Supplement: Matched Placebo

INTERVENTIONS:
Dietary Supplement: Lemon Balm Supplement — Oral 200 mg Lemon Balm supplement tablet Twice a day for three-weeks
  Arms: Supplement Group
Dietary Supplement: Matched Placebo — Matched placebo tablet Twice a day for three-weeks
  Arms: Control group

SUMMARY:
This study is aimed to investigate if Lemon Balm Extract supplementation is beneficial for the relief of stress, depression and anxiety in healthy adults.

DETAILED DESCRIPTION:
Lemon balm (Botanical name: Melissa officinalis L.) is a herbal plant belongs to the Lamiaceae (mint) family, and currently of wide scientific interest as possible adjuvant for calming effect. Lemon balm is one of the most popular and widely used medicinal herbs in central and southern Europe, the Mediterranean region, and west Asia. The European Scientific Cooperative on Phytotherapy (ESCOP) recommends the use of lemon balm to relieve of mild symptoms of anxiety, including mental stress, restlessness, and irritability. Historically, Lemon balm has been widely used in Asian traditional medicine as a sedative to treat many psychiatric disorders, such as stress, depression, anxiety, and insomnia. Lemon balm has shown anti-depressant, anxiolytic, and anti-insomnia effects both in human clinical trials and in animal model studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, aged 18 - 65 years
* Individuals suffering from moderate degree of depression, anxiety, and stress with DASS scores ≥14, ≥10, and ≥19, respectively, or individual with sleep problems with Pittsburgh Sleep Quality Index (PSQI) score ≥5.
* Willing to participate in the study

Exclusion Criteria:

* Current use of prescribed medication or supplements for neuropsychiatric and sleep disorders
* Known history of neuropsychiatric or sleep disorders
* Current use or history of illicit substances misuse
* History of any allergic reactions to ingredients of the Lemon Balm Extract
* Hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90, or other cardiovascular disease
* Hyperthyroidism or Diabetes mellitus or cancer
* Use of blood thinners like Coumadin (warfarin) or Plavix (clopidogrel), Glaucoma medications like Travatan (travoprost), Chemotherapy drugs like tamoxifen and Camptosar (irinotecan)
* Severe medical problem, which in the opinion of the investigator would pose a safety risk to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in the level of depression | 3 weeks
  Improvement in the Depression score in the Depression Anxiety and Stress Scale (DASS)
Changes in the level of anxiety | 3 weeks
  Improvement in the Anxiety score in the Depression Anxiety and Stress Scale (DASS)
Changes in the level of stress | 3 weeks
  Improvement in the Stress score in the Depression Anxiety and Stress Scale (DASS)
Changes in sleep quality | 3 weeks
  Improvement in the Pittsburgh Sleep Quality Index (PSQI) scale score

SECONDARY OUTCOMES:
Changes in mental wellbeing | 3 weeks
  Improvement in the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) score
Changes in Positive and Negative Emotional Feelings | 3 weeks
  Improvement in the Positive and Negative Affect Scale (PANAS) score
Changes in the Quality of Life (QoL) | 3 weeks
  Improvement in the WHO QOL-BREF scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Ayub Teaching Hospital, Abbottābād, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alijaniha F, Naseri M, Afsharypuor S, Fallahi F, Noorbala A, Mosaddegh M, Faghihzadeh S, Sadrai S. Heart palpitation relief with Melissa officinalis leaf extract: double blind, randomized, placebo controlled trial of efficacy and safety. J Ethnopharmacol. 2015 Apr 22;164:378-84. doi: 10.1016/j.jep.2015.02.007. Epub 2015 Feb 11. PMID 25680840
- [Background] Araj-Khodaei M, Noorbala AA, Yarani R, Emadi F, Emaratkar E, Faghihzadeh S, Parsian Z, Alijaniha F, Kamalinejad M, Naseri M. A double-blind, randomized pilot study for comparison of Melissa officinalis L. and Lavandula angustifolia Mill. with Fluoxetine for the treatment of depression. BMC Complement Med Ther. 2020 Jul 3;20(1):207. doi: 10.1186/s12906-020-03003-5. PMID 32620104
- [Background] Ballard CG, O'Brien JT, Reichelt K, Perry EK. Aromatherapy as a safe and effective treatment for the management of agitation in severe dementia: the results of a double-blind, placebo-controlled trial with Melissa. J Clin Psychiatry. 2002 Jul;63(7):553-8. doi: 10.4088/jcp.v63n0703. PMID 12143909
- [Background] Emamghoreishi, M. and M.S. Talebianpour, Antidepressant effect of Melissa officinalis in the forced swimming test. DARU, 2009. 17: p. 42-47
- [Background] Haybar H, Javid AZ, Haghighizadeh MH, Valizadeh E, Mohaghegh SM, Mohammadzadeh A. The effects of Melissa officinalis supplementation on depression, anxiety, stress, and sleep disorder in patients with chronic stable angina. Clin Nutr ESPEN. 2018 Aug;26:47-52. doi: 10.1016/j.clnesp.2018.04.015. Epub 2018 May 19. PMID 29908682
- [Background] Heydari N, Dehghani M, Emamghoreishi M, Akbarzadeh M. Effect of Melissa officinalis capsule on the mental health of female adolescents with premenstrual syndrome: a clinical trial study. Int J Adolesc Med Health. 2018 Jan 25;31(3):/j/ijamh.2019.31.issue-3/ijamh-2017-0015/ijamh-2017-0015.xml. doi: 10.1515/ijamh-2017-0015. PMID 29369810
- [Background] Kennedy DO, Little W, Haskell CF, Scholey AB. Anxiolytic effects of a combination of Melissa officinalis and Valeriana officinalis during laboratory induced stress. Phytother Res. 2006 Feb;20(2):96-102. doi: 10.1002/ptr.1787. PMID 16444660
- [Background] Kennedy DO, Little W, Scholey AB. Attenuation of laboratory-induced stress in humans after acute administration of Melissa officinalis (Lemon Balm). Psychosom Med. 2004 Jul-Aug;66(4):607-13. doi: 10.1097/01.psy.0000132877.72833.71. PMID 15272110
- [Background] Kennedy DO, Scholey AB, Tildesley NT, Perry EK, Wesnes KA. Modulation of mood and cognitive performance following acute administration of Melissa officinalis (lemon balm). Pharmacol Biochem Behav. 2002 Jul;72(4):953-64. doi: 10.1016/s0091-3057(02)00777-3. PMID 12062586
- [Background] Kennedy DO, Wake G, Savelev S, Tildesley NT, Perry EK, Wesnes KA, Scholey AB. Modulation of mood and cognitive performance following acute administration of single doses of Melissa officinalis (Lemon balm) with human CNS nicotinic and muscarinic receptor-binding properties. Neuropsychopharmacology. 2003 Oct;28(10):1871-81. doi: 10.1038/sj.npp.1300230. PMID 12888775
- [Background] Ranjbar M, Firoozabadi A, Salehi A, Ghorbanifar Z, Zarshenas MM, Sadeghniiat-Haghighi K, Rezaeizadeh H. Effects of Herbal combination (Melissa officinalis L. and Nepeta menthoides Boiss. & Buhse) on insomnia severity, anxiety and depression in insomniacs: Randomized placebo controlled trial. Integr Med Res. 2018 Dec;7(4):328-332. doi: 10.1016/j.imr.2018.08.001. Epub 2018 Aug 10. PMID 30591886
- [Background] Ranjbar M, Salehi A, Rezaeizadeh H, Zarshenas MM, Sadeghniiat-Haghighi K, Mirabzadeh M, Firoozabadi A. Efficacy of a Combination of Melissa officinalis L. and Nepeta Menthoides Boiss. & Buhse on Insomnia: A Triple-Blind, Randomized Placebo-Controlled Clinical Trial. J Altern Complement Med. 2018 May 9. doi: 10.1089/acm.2017.0153. Online ahead of print. PMID 29741926
- [Background] Shirazi M, Jalalian MN, Abed M, Ghaemi M. The Effectiveness of Melissa Officinalis L. versus Citalopram on Quality of Life of Menopausal Women with Sleep Disorder: A Randomized Double-Blind Clinical Trial. Rev Bras Ginecol Obstet. 2021 Feb;43(2):126-130. doi: 10.1055/s-0040-1721857. Epub 2021 Jan 19. PMID 33465795
- [Background] Soltanpour, A., et al., Effects of Melissa officinalis on anxiety and sleep quality in patients undergoing coronary artery bypass surgery: A double-blind randomized placebo controlled trial. European Journal of Integrative Medicine, 2019. 28: p. 27-32
- [Result] Cases J, Ibarra A, Feuillere N, Roller M, Sukkar SG. Pilot trial of Melissa officinalis L. leaf extract in the treatment of volunteers suffering from mild-to-moderate anxiety disorders and sleep disturbances. Med J Nutrition Metab. 2011 Dec;4(3):211-218. doi: 10.1007/s12349-010-0045-4. Epub 2010 Dec 17. PMID 22207903
- [Derived] Bano A, Hepsomali P, Rabbani F, Farooq U, Kanwal A, Saleem A, Bugti AA, Khan AA, Khalid Z, Bugti M, Mureed S, Khan S, Ujjan ID, Sahin S, Kara M, Khan A. The possible "calming effect" of subchronic supplementation of a standardised phospholipid carrier-based Melissa officinalis L. extract in healthy adults with emotional distress and poor sleep conditions: results from a prospective, randomised, double-blinded, placebo-controlled clinical trial. Front Pharmacol. 2023 Oct 19;14:1250560. doi: 10.3389/fphar.2023.1250560. eCollection 2023. PMID 37927585